CLINICAL TRIAL: NCT06217757
Title: Phase I Study of Low-Dose Radiotherapy Plus Chemotherapy and Sugemalimab and Olaparib for First-Line Treatment of SLFN-11 Positive Extensive Stage Small Cell Lung Cancer
Brief Title: Safety and Tolerability of LDRT+Sugemalimab+Chemotherapy+Olaparib for First-Line Treatment of SLFN-11 Positive ES-SCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Chief of Thoracic Cancer Ward, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCS-Lung01
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer; Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Radiotherapy; Etoposide; Cisplatin; sugemalimab; olaparib; ADP Ribose Transferases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low-dose radiotherapy combined with sugemalimab, olaparib, etoposide and cisplatin (Experimental): Participants will receive the following treatment regimens: LDRT cisplatin + etoposide + sugemalimab+olaparib. Induction treatment will be administered on a 21-day cycle for four cycles. LDRT will be conducted from Day 1 - Day 5 in the first cycle. Following the induction phase, participants will continue maintenance therapy with sugemalimab and olaparib. Participants will be treated until loss of clinical benefit, or unaccepted toxicity, or withdrawal of consent, or death (whichever occurs first).
  Interventions: Radiation: Low-dose radiotherapy; Drug: Etoposide; Drug: Cisplatin; Drug: Sugemalimab; Drug: Olaparib

INTERVENTIONS:
Radiation: Low-dose radiotherapy — The LDRT deals with primary tumour in a 15 Gy of 5fractions over five days, starting from Day 1 in the first cycle.
  Other Names: LDRT
Drug: Etoposide — Etoposide will be administered intravenously at a dose of 100 mg/m^2 on Days 1, 2 and 3 of each 21-day cycle during the induction phase (Cycles 1-4).
  Other Names: One of the standard chemotherapy regimens
Drug: Cisplatin — Cisplatin will be administered as intravenous infusion at a dose of 25 mg/m^2 on Days 1, 2 and 3 of each 21-day cycle during the induction phase (Cycles 1-4).
  Other Names: One of the standard chemotherapy regimens
Drug: Sugemalimab — Sugemalimab will be administered by intravenous infusion at a dose of 1200mg on Day 1 of each 21-day cycle for a maximum of 2 years or progressive disease or intolerable toxicity.
  Other Names: Programmed Death Ligand-1 (PD-L1) Inhibitor
Drug: Olaparib — Olaparib will be administered orally at a dose of 150mg qod Day 1,3,5,7 or 150 mg qd/150 mg bid/300mg in the morning and 150mg in the evening/300 mg bid on Day 1-7 of each 21-day cycle for a maximum of 2 years or progressive disease or intolerable toxicity.
  Other Names: poly ADP-ribose polymerase (PARP) inhibitor

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of low-dose radiotherapy (LDRT) combined with sugemalimab, olaparib, chemotherapy in the first-line treatment of SLFN-11 positive extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
This study consists of dose escalation and dose expansion in China. Subjects who fulfil all the inclusion criteria and none of the exclusion criteria will be enrolled and receive treatment with Sugemalimab, Etoposide/Cisplatin Chemotherapy and Olaparib for 4 cycles with LDRT in the first cycle. Sugemalimab in combination with olaparib will be administered for maintenance therapy after 4 cycles. Sugemalimab will be administered at a dose of 1200 mg every 3 weeks (Q3W) in the first day of every cycle. The LDRT deals with primary tumour in a 15 Gy of 5 fractions over five days, starting from day 1 in the first cycle. Dose of olaparib will identify by assessed recommended dose for expansion (RDE) in dose escalation stage.A dose expansion stage will be conducted after dose escalation. The primary endpoint is safety.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years old and less than or equal to (≤) 75 years old
2. Histologically or cytologically confirmed ES-SCLC
3. No prior treatment for ES-SCLC
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Five white slides (unstained paraffin sections) were available for immunohistochemical SLFN-11 detection and SLFN-11 was positive
6. Extensive clinical stage. American Joint Committee on Cancer (AJCC) 8th edition Stage IV with lesions exceeding one side of the chest and including malignant pleural and pericardial effusions or hematogenous metastases (any T, any N, M1a/b/c); or T3-4 due to multiple nodules in the lung or tumor/nodule size too large to be included in a T3-4 disease within a tolerable radiotherapy schedule
7. The subjects were considered suitable for combining etoposide with cisplatin chemotherapy and low-dose radiotherapy as first-line treatment for extensive -stage small cell lung cancer
8. Have measurable lesions as defined by RECIST1.1, with at least one lesion (never previously treated with radiation) of ≥10 mm longest diameter accurately measured by computed tomography (CT) or magnetic resonance imaging (MRI) at baseline (except for lymph nodes, which must have a short axis of ≥15 mm) and the lesion is suitable for repeat and accurate measurements
9. Patients with brain metastases must be asymptomatic or stable on steroids and anticonvulsants for at least 1 month prior to study treatment. Participants with suspected brain metastases during screening should have a CT/MRI of the brain prior to study
10. No previous treatment with immune checkpoint inhibitors and PARP inhibitors, including but not limited to other anti-PD-1, anti-PD-L1 and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, with the exception of therapeutic anti-tumor vaccines. No prior chemotherapy or radiation therapy to the chest lesion
11. Weight over 30 Kg
12. Life expectancy ≥ 12 weeks
13. Have adequate organ and bone marrow functional reserve and normal major organ function
14. Patients were compliant, voluntarily enrolled in the study and signed an informed consent form
15. For women or men with childbearing potential: use effective contraception to avoid conception or embryonic drug exposure during treatment and for 5 months after the last dose of sugemalimab and for 6 months after the last dose of cisplatin or etoposide. Female subjects are prohibited from donating eggs during this period and males are prohibited from donating sperm during this period

Exclusion Criteria:

1. Histopathologic or cytopathologic diagnosis of mixed small cell lung cancer or non-small cell lung cancer
2. Limited stage small cell lung cancer
3. Combination of poorly controlled malignant pleural or pericardial effusions requiring continuous drainage
4. Presence of active or symptomatic brain metastases or Leptomeningeal metastases
5. Prior systemic antitumor therapy (chemotherapy, targeted agents such as PARP inhibitors) or immune checkpoint inhibitors for SCLC
6. Presence of active, unstable systemic disease such as active infection, autoimmune disease, inflammatory disease (uncontrolled hypertension, heart failure (NYHA classification >= Class II), unstable angina, acute coronary syndrome, severe arrhythmia, severe hepatic, renal or metabolic disease, human immunodeficiency virus (HIV) immunodeficiency virus (HIV) infected patients
7. Previous allogeneic stem cell or solid organ transplantation
8. Patients with prior interstitial lung disease, drug-induced interstitial lung disease, or active interstitial pneumonia requiring systemic glucocorticoid or immunosuppressive therapy; Patients with pulmonary interstitial fibrosis or active pulmonary tuberculosis
9. Severe infection within 4 weeks prior to the start of study treatment, including but not limited to hospitalization for infection, bacteremia, or severe pneumonia
10. Received therapeutic oral or intravenous infusion of antibiotics within 2 weeks prior to the start of study treatment
11. Been diagnosed or treated for another malignancy (excluding resected basal cell carcinoma of the skin or other carcinoma in situ) within 5 years prior to randomization to this study
12. For pregnant or lactating females or male or female subjects of reproductive potential who refuse to use effective contraception during treatment and within 5 months of the last dose of sugemalimab and within 6 months of the last dose of cisplatin or etoposide
13. Allergic to the study drug or its components
14. The investigator believes that the patients may not be able to complete the study or comply with the requirements of the study
15. Inadequate bone marrow function and vital organ function reserve
16. Concurrent participation in another clinical study, unless it is an observational (non-interventional) clinical study or a follow-up phase of an interventional study, excluding patients who have received any other experimental drug within 28 days prior to the start of study treatment
17. Patients who are not suitable for etoposide-cisplatin chemotherapy, sugemalimab or olaparib
18. History of thoracic radiotherapy or plan to receive intensive thoracic radiotherapy prior to systemic therapy. External chest radiotherapy for palliative purposes (e.g., bone metastases) is allowed, but must be completed prior to the first administration of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
RDE | 3 weeks after initiation of treatment.
  To determine the RDE of olaparib in subjects with Extensive Stage-SCLC when combined with low-Dose Radiotherapy, chemotherapy and sugemalimab.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Baseline up to approximately 24 months
  The time from the date of first dosing of sugemalimab to the first appearance of objective disease progression (according to RECIST1.1) or death from any cause (if it occurs before disease progression).
PFS Rate at 6 Months and 1 Year | Baseline up to 1 year
  PFS rate at 6 months and 1 year, defined as the proportion of patients who have not experienced disease progression or death from any cause at 6 months and 1 year separately, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST1.1).
Overall Survival (OS) | Baseline up to approximately 24 months
  OS, defined as the time from initiation of study treatment to death from any cause.
OS Rate at 1 Year, 1.5 Years and 2 Years | Baseline to 2 years or death, whichever occurs first.
  OS rate at 1 year, 1.5 years and 2 years, defined as the proportion of patients who have not experienced death from any cause at 1 year ,1.5 years and 2 years.
Objective response rate (ORR) | Baseline to 2 years
  According to the evaluation criteria of RECIST1.1

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaczorowski M, Ylaya K, Chlopek M, Taniyama D, Pommier Y, Lasota J, Miettinen M. Immunohistochemical Evaluation of Schlafen 11 (SLFN11) Expression in Cancer in the Search of Biomarker-Informed Treatment Targets: A Study of 127 Entities Represented by 6658 Tumors. Am J Surg Pathol. 2024 Dec 1;48(12):1512-1521. doi: 10.1097/PAS.0000000000002299. Epub 2024 Aug 26. PMID 39185596